CLINICAL TRIAL: NCT07386158
Title: Phase II Single-arm Clinical Study of the Efficacy and Safety of Pucotenlimab in Combination With Vorolanib Neoadjuvant Therapy for Patients With High-risk Renal Carcinoma Indicating Partial Nephrectomy
Brief Title: Pucotenlimab Combination With Vorolanib as Neoadjuvant Therapy for ccRCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-041-01
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: Vorolanib; Clear Cell Renal Cell Carcinoma (ccRCC); Neoadjuvant Therapy
Keywords: Vorolanib; Clear Cell Renal Cell Carcinoma (ccRCC); Neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — vorolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pucotenlimab combination with Vorolanib as neoadjuvant therapy (Experimental): Vorolanib Treatment Vorolanib 200mg orally once daily, with or without food.Intravenous Infusion of Pucotenlimab(Injection) Infuse Pucotenlimab at a dose of 200mg intravenously every three weeks, constituting one treatment cycle, the maximum duration of treatment should not exceed 4 cycles.Perform imaging evaluation after 2 cycles, including renal CT plain scan+enhancement, measurement of tumor volume, and evaluation of ORR. If PD is detected in the first imaging assessment, the study will be terminated. According to the current diagnosis and treatment routine, communicate with the patient about the follow-up treatment plan:Radical nephrectomy; Utilization of other targeted therapies; Combination targeted therapy with immunotherapy. If the tumor shrinks significantly and the surgeon evaluates that partial nephrectomy can be safely performed, drug therapy should be stopped and partial nephrectomy should be performed; otherwise, continue treatment to 4 cycles before surgery.
  Interventions: Drug: Pucotenlimab combination with Vorolanib

INTERVENTIONS:
Drug: Pucotenlimab combination with Vorolanib — 3.7.1 Vorolanib Vorolanib 200mg PO QD, taken with or without food. 3.7.2 Pucotenlimab Intravenous infusion of 200mg of Pucotenlimab (injection), once every 3 weeks, as one treatment cycle.

SUMMARY:
Through the neoadjuvant treatment with a combination of Pucotenlimab and Vorolanib, it enabled the successful and safe implementation of partial nephrectomy in patients with localized renal cancer, who had indications for nephron-sparing surgery but faced considerable difficulty in preserving the kidney (T1b with an endophytic component ≥75% or T2)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form (ICF).
2. Age at the time of enrollment is between 18 years old and 85 years old, regardless of gender.
3. The physical fitness score of the Eastern Cooperative Oncology Group (ECOG) in the United States is 0 or 1.
4. Expected survival period ≥ 3 months.
5. Preoperative biopsy pathology confirms renal clear cell carcinoma or renal cell carcinoma mainly composed of clear cell carcinoma
6. ECOG score 0 or 1
7. The patient is willing to undergo kidney preservation surgery
8. Preoperative assessment of healthy kidney GFR<60 ml/min through renal dynamic imaging
9. There are indications for kidney preservation surgery, but the surgery is difficult [① 4-7cm tumor located at the renal hilum or endogenous ≥ 75% (T1bN0M0); ② Tumors larger than 7cm (T2N0M0)] 9. There should be at least one measurable lesion (according to mRECIST v1.1 criteria) that is suitable for repeated and accurate measurements.
10. Good organ function, laboratory test results during the screening period meet the following criteria:

<!-- -->

1. Hematology (no blood components or cell growth factors are allowed to support treatment within 2 weeks before starting treatment):

   a. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1500/mm3); b. Platelet count (PLT) ≥ 100 × 109/L (100000/mm3); c. Hemoglobin (HB) ≥ 90 g/L;
2. Liver:

   1. Serum total bilirubin (TBIL) ≤ 1.5 × ULN;
   2. Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 × ULN; For subjects with liver metastasis, AST and ALT ≤ 5 × ULN
   3. Serum albumin (ALB) ≥ 28g/L
3. Coagulation function:

   International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN 11. The subjects are willing and able to comply with the scheduled visits, treatment plans, laboratory tests, and other requirements of the study.

   Exclusion Criteria:

   • Renal vein cancer thrombus

   • Diffuse tumor growth, with no clear boundary from normal renal parenchyma

   • General poor condition, anesthesia assessment cannot tolerate general anesthesia surgery

   • Have serious cardiovascular and cerebrovascular diseases, uncontrollable

   • hypertension and diabetes

   • Patients who have long-term use of immunosuppressants after organ transplantation

   • Patients who are currently using immunosuppressive drugs

   • Patients with clear infection or fever

   • Patients with T-cell lymphoma and myeloma

   • Patients who have concurrent malignant tumors, are currently undergoing treatment for other benign or malignant tumors, or have a history of other malignant tumors within the past six months

   • Metastatic renal cell carcinoma.

   • Received Chinese herbal medicine or immunomodulatory drugs with anti-tumor indications within 14 days prior to the first use of the investigational drug

   • Perform systematic treatment (including thymosin, interferon, interleukin, except for local use to control pleural effusion).

   • Suffering from active or potentially recurrent autoimmune diseases, except for vitiligo, hair loss, psoriasis, or eczema that do not require systemic treatment; Hypothyroidism caused by autoimmune thyroiditis only requires stable doses of hormone replacement therapy; Type I diabetes requiring only a stable dose of insulin replacement therapy.

   • Simultaneously enrolled in another clinical study, unless it is an observational, non interventional clinical study or a follow-up period of an interventional study.

   Known history of mental illness, drug abuse, alcoholism, or drug use.
   * Pregnant or lactating women.
   * Any past or current illness, treatment, or laboratory test abnormalities may confuse the research results, affect the full participation of the subjects in the study, or participation in the study may not be in the best interests of the subjects.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) based on RECIST 1.1 criteria. | Evaluation at the end of Cycle 2 or Cycle 4 (each cycle is 21 days) of Pucotenlimab treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No